CLINICAL TRIAL: NCT01352533
Title: A Randomized Prospective Trial of 2-Octyl Cyanoacrylate (Derma-Bond) Tissue Adhesive Versus Running Subcuticular Suture Combined With Tissue Adhesive Versus Epidermal Sutures in Dermatologic Surgery Procedures of the Head and Neck
Brief Title: Closure Techniques and Scar Appearance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Associate Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU38040
Record Dates: First submitted 2011-04-29; First posted 2011-05-12 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Wound Closure Techniques
MeSH Terms: interventions — Tissue Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Running polypropylene closure (Active Comparator): Half of every linear wound will be closed with running polypropylene sutures. This technique is Standard of Care.
  Interventions: Procedure: Running polypropylene closure
- Tissue Adhesive (Derma-Bond) (Experimental): The experimental half of the wound will be randomized to receive closure with tissue adhesive alone.
  Interventions: Procedure: Tissue Adhesive (Derma-Bond)
- Subcuticular polyglactin-910 combined with tissue adhesive (Experimental): The experimental half of the wound will be randomized to receive closure with running subcuticular polyglactin-910 combined with tissue adhesive.
  Interventions: Procedure: Subcuticular polyglactin-910 combined with tissue adhesive

INTERVENTIONS:
Procedure: Running polypropylene closure — Half of every wound will be closed with Standard of Care running polypropylene sutures
  Arms: Running polypropylene closure
Procedure: Tissue Adhesive (Derma-Bond) — Approximately half of wounds will be randomized to be closed with tissue adhesive.
  Arms: Tissue Adhesive (Derma-Bond)
Procedure: Subcuticular polyglactin-910 combined with tissue adhesive — Approximately half of the experimental wounds will be randomized to be closed with a combination of subcuticular polyglactin-910 and tissue adhesive.
  Arms: Subcuticular polyglactin-910 combined with tissue adhesive

SUMMARY:
The goal of this study is to assess whether wound closure with skin adhesive or running stitches combined with skin adhesive will be superior to standard wound sutures. This is a split-wound study that will compare two methods of skin closure within one standard closure technique, thereby providing an internal control of running stitches within each wound. The investigators plan to measure outcomes by assessing for scar appearance, the incidence of wound opening, scar elasticity and subject satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Linear closures on the head and neck, at least 3cm in length
* The subjects are in good health
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.

Exclusion Criteria:

* Under 18 years of age
* Pregnancy or Lactation
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness
* Defects on the scalp

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 10 day/3 weeks and 3 months
  The primary outcome measure of this study will be wound healing. This outcome will be assessed by the blinded observers, subject ratings and Cutometer measurements of scar elasticity. Two double-blinded dermatologists will be asked to rate the scars according to the objective scar scales at the 10 day/ 3 week and 3 month follow-up exams.

SECONDARY OUTCOMES:
Dehiscence | 10 days/3 weeks and 3 months
  The rate of dehiscence observed will be noted and recorded by the treating physicians.
Subject Satisfaction | 10 days/3 weeks and 3 months
  The subjects will fill out the VAS to evaluate their overall assessment of their scar, any associated pruritus and pain. The subjects will also fill out a Subject Satisfaction Survey to evaluate subject preference for closure.
Adverse Events | 10 days/3 weeks and 3 months
  The treating physicians will note occurrence and extent of any adverse events associated with either type of epidermal closure.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University